CLINICAL TRIAL: NCT01447394
Title: A Double-Blinded Randomized Control Study Evaluating the Efficacy and Safety of Pegylated Lambda Interferon Compared to Pegylated Alfa-2a Interferon, Each in Combination With Ribavirin, in the Treatment of Naive Genotype 1 or 4 Chronic Hepatitis C Subjects
Brief Title: Safety and Efficacy Study of Pegylated Interferon Lambda Versus Pegylated Interferon Alfa, Plus Ribavirin in Subjects With Hepatitis C
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI452-013; 2011-003748-31 (EudraCT Number)
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C Virus (HCV)
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Pegylated Interferon Lambda + Ribavirin (Experimental)
  Interventions: Biological: Pegylated Interferon Lambda; Drug: Ribavirin
- Arm 2: Pegylated Interferon Alfa-2a + Ribavirin (Active Comparator)
  Interventions: Biological: Pegylated Interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Biological: Pegylated Interferon Lambda — Syringe, Subcutaneous, 180 μg, Once weekly, 48 weeks
  Other Names: BMS-914143
  Arms: Arm 1: Pegylated Interferon Lambda + Ribavirin
Biological: Pegylated Interferon Alfa-2a — Syringe, Subcutaneous, 180 μg, Once weekly, 48 weeks
  Other Names: Pegasys
  Arms: Arm 2: Pegylated Interferon Alfa-2a + Ribavirin
Drug: Ribavirin — Tablets, Oral, 1000 or 1200 mg based on weight, Twice daily, 48 weeks
  Other Names: Ribasphere

SUMMARY:
The purpose of this study is to determine if 48 weeks of therapy with Pegylated Interferon Lambda plus Ribavirin is effective and safe for a treatment of chronic hepatitis C (CHC) compared to therapy with Pegylated Interferon Alfa-2a plus Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C, Genotype 1 or 4
* HCV Ribonucleic acid (RNA) ≥ 100,000 IU/mL at screening
* Liver biopsy documenting no cirrhosis (within prior 2 years) or cirrhosis (from any time prior to randomization). Where approved for staging of liver disease, non-invasive imaging may be used to assess the extent of liver disease. Subjects with compensated cirrhosis can enroll and will be capped at 10%
* Naive to prior anti-HCV therapy

Exclusion Criteria:

* Infected with HCV other than Genotype 1 or 4
* Positive Hepatitis B surface antigen (HBsAg), or Human immunodeficiency virus-1 (HIV-1)/HIV-2 antibody or hepatitis D virus (HDV) at screening
* Evidence of liver disease other than HCV
* Active substance abuse
* Use of hematologic growth factors within 90 days prior to study randomization
* Evidence of decompensated cirrhosis based on radiologic criteria or biopsy results and clinical criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Lambda + Ribavirin (RBV) compared to Alfa + RBV in achieving a sustained virological response | At follow-up Week 24 (SVR24) following 48 weeks of treatment
The safety of Lambda + RBV compared to Alfa + RBV in reducing cytopenic abnormalities | From Day 1 to end of Week 48 on-treatment

SECONDARY OUTCOMES:
Proportion of interferon-associated symptoms: a) Flu-like symptoms b) Musculoskeletal symptoms c) Neurologic symptoms d) Psychiatric symptoms e) Constitutional symptoms | From Day 1 to end of Week 48 on-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (80):
- United States (3):
  - Local Institution, San Diego, California
  - Local Institution, Rochester, New York
  - Local Institution, Houston, Texas
- Canada (2):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Vaughan, Ontario
- Local Institution, Hong Kong, Hong Kong, China
- Colombia (3):
  - Local Institution, Bogotá
  - Local Institution, Cali
  - Local Institution, Medellín
- Czechia (3):
  - Local Institution, Hradec Králové
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
- Egypt (2):
  - Local Institution, Shebin Elkom, Monufia Governorate
  - Local Institution, Cairo
- Hong Kong (2):
  - Local Institution, Lai Chi Kok
  - Local Institution, Tai Po
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Miskolc
- India (6):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Coimbatore
  - Local Institution, Gūrgaon
  - Local Institution, Ludhiana
  - Local Institution, Nagpur
  - Local Institution, New Delhi
- Local Institution, Dublin, Dublin, Ireland
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
- Poland (15):
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Chorzów
  - Local Institution, Czeladź
  - Local Institution, Kielce
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Olsztyn
  - Local Institution, Puławy
  - Local Institution, Racibórz
  - Local Institution, Sosnowiec
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Zielona Góra
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Iași
  - Local Institution, Timișoara
- Russia (12):
  - Local Institution, Yoshkar-Ola, Mariy-El Republic
  - Local Institution, Kaluga
  - Local Institution, Lipetsk
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Poselok Noviy
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Saratov
  - Local Institution, Smolensk
  - Local Institution, Tolyatti
  - Local Institution, Volgograd
- Local Institution, Singapore, Singapore
- South Korea (5):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Incheon
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (3):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Taiwan (5):
  - Local Institution, Taipei, Taiwan
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
- Turkey (Türkiye) (5):
  - Local Institution, Ankara
  - Local Institution, Bornova Izmir
  - Local Institution, Diyarbakır
  - Local Institution, Istanbul
  - Local Institution, Trabzon
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Edinburgh, Midlothian
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx